CLINICAL TRIAL: NCT04389229
Title: Protocol Title: An Open Label, Multi-centre Phase 1/2a Study of Modified and Unmodified Autologous Tumour Infiltrating Lymphocytes (TIL) in Patients With Platinum-resistant Ovarian Cancer
Brief Title: OVSTAR TIL Trial (OVarian Cancer Co-STimulatory Antigen Receptor TIL Trial)
Acronym: OVSTAR
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Immetacyte Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMM-2019T-01-OC; 2019-000106-30 (EudraCT Number)
Record Dates: First submitted 2020-01-22; First posted 2020-05-15 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Ovarian Cancer Metastatic
MeSH Terms: interventions — Cyclophosphamide; fludarabine; Interleukin-2; aldesleukin

STUDY DESIGN:
Intervention Model Description: This study has two cohorts which will open sequentially. This is not a randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UTIL-01 (Experimental): Single dose autologous unmodified tumour infiltrating lymphocytes
  Interventions: Drug: cyclophosphamide; Drug: fludarabine; Drug: IL-2 (Proleukin); Genetic: Unmodified Tumour Infiltrating Lymphocytes (UTIL-01)
- CoTIL-01 (Experimental): Single dose autologous gene modified tumour infiltrating lymphocytes
  Interventions: Drug: cyclophosphamide; Drug: fludarabine; Drug: IL-2 (Proleukin); Genetic: Gene modified Tumour Infiltrating Lymphocytes (CoTIL-01)

INTERVENTIONS:
Drug: cyclophosphamide — 600mg/m2/day for 3 days ( on day -5, -4, -3)
Drug: fludarabine — 30mg/m2/day for 3 days ( on day -5, -4, -3)
Drug: IL-2 (Proleukin) — Subcutaneous injections at a fixed dose of 18 million units once a day following TIL infusion
Genetic: Unmodified Tumour Infiltrating Lymphocytes (UTIL-01) — Single dose at 5 x 10^9 - 5 x 10^10
  Other Names: TIL
  Arms: UTIL-01
Genetic: Gene modified Tumour Infiltrating Lymphocytes (CoTIL-01) — Single dose at 2 x10^9 (+/- 20%) (engineered TIL)
  Other Names: engineeredTIL
  Arms: CoTIL-01

SUMMARY:
An open label, multi-centre Phase 1/2a study of modified and unmodified autologous Tumour Infiltrating Lymphocytes (TIL) in patients with platinum-resistant ovarian cancer. The purpose of this phase I/II study is to evaluate the feasibility and safety of both standard unmodified TIL (UTIL-01) and TIL engineered to express the co-stimulatory receptor CoStAR (CoTIL-01) in platinum resistant ovarian cancer.

DETAILED DESCRIPTION:
This is a single-arm Phase 1/2a study of unmodified (UTIL-01) and gene modified (CoTIL-01) adoptive TIL therapy which will enrol sequentially. A total of 8 patients will be recruited to the UTIL-01 cohort to receive autologous standard unmodified TIL (phase 2). Up to 14 patients will receive autologous gene engineered TIL(CoTIL-1) in a dose escalation design (Phase 1/2a). Once patients have met all the pre-screening inclusion criteria, and that sponsor has confirmed a successful TIL harvest, a request to manufacture will be sent to the Sponsor to initiate TIL production. Manufacturing and quality control assessment is anticipated to take approximately 6 weeks. During this time, patients may receive standard of care chemotherapy (bridging chemotherapy) as deemed appropriate by the treating oncology team. Patients will proceed to the main trial after completion of bridging chemotherapy. Once the TIL product is certified for release, and that patient has consented to the main trial and has completed main trial screening assessments, study treatment can be scheduled.

Patients will receive non-myeloablative lymphodepleting pre-conditioning chemotherapy with cyclophosphamide 600mg/m2/day and fludarabine 30mg/m2/day on Day -5, -4 and -3. Chemotherapy will aim to be delivered as an outpatient, but patients can be admitted if clinically needed. Patients will be required to maintain oral hydration of >2 litres per day. If this is felt to be difficult to achieve then the patient will be admitted for IV fluids. Patients will be admitted for TIL infusion on Day 0. The TIL infusion will be administered at least 36 hours after last dose of chemotherapy. The cells will only be thawed once an Investigator has made a positive decision to go ahead with infusion and confirmed this in writing. TIL infusion may be delayed for up to 7 days for clinical reasons or for issues regarding the cell specification. This decision must be made before final preparation for infusion. Following TIL infusion, patients will commence subcutaneous interleukin-2 at a fixed dose of 18 million units once a day. Patients must remain an inpatient for the duration of IL-2 treatment for a minimum of 7 days post TIL infusion. Recruitment to the study will occur over approximately 24-month period. Recruitment to CoTIL-01 will commence after UTIL-01. Patients will be followed up in the study for 24 months post TIL infusion.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for Pre-Screening Phase

Patients are eligible to be included in the pre-screening phase of the study only if all of the following criteria apply:

1. Women with histologically confirmed recurrent metastatic platinum-resistant high-grade serous ovarian cancer (HGSOC) (platinum resistant defined as progressing within 6 months of last platinum-containing combination chemotherapy. Patients must have received at least 1 line of prior platinum-containing combination chemotherapy and have completed at least 4 cycles of this treatment).
2. Expected to fulfil all entry criteria for OVSTAR Main Study
3. Written informed consent to Pre-Screening
4. Measurable disease by Response Evaluation Criteria in Solid Tumours 1.1
5. Have disease suitable for fresh TIL harvesting from tumour biopsies (only applicable to patients who are not participants of Sponsor's Tumour Collection Programme, PRIME)
6. Medically suitable for a general anaesthetic and surgical biopsy (only applicable to patients who are not participants of Sponsor's Tumour Collection Programme, PRIME)
7. Women of child bearing potential must be willing to practise a highly effective method of birth control once consented to pre-screening
8. World Health Organisation (WHO) Performance Status of 0 or 1 (Appendix 3)
9. Age equal to or greater than 18 years
10. Life expectancy > 6 months
11. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the Pre-Screening or Main Study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
12. Seronegative for HIV antibody, Hep B antigen, Hep C antibody and syphilis
13. Haematological and biochemical indices

Exclusion Criteria:

* Exclusion for Pre-Screening Phase

Patients will not be invited to participate in Pre-Screening if any of the following criteria apply:

1. History of a previous malignancy at another site, unless followed for >2 years with no sign of recurrent disease (local completely excised cutaneous basal cell, squamous cell carcinoma or in situ carcinoma will be allowed).
2. Patients receiving chemotherapy, targeted therapy, immunotherapy or systemic steroids including steroid doses >10mg/day of prednisolone (or equivalent) during the previous four weeks prior to TIL harvesting. Patients who require such therapies intermittently due to pre-existing disorders are also excluded.
3. Evidence of any active significant infection.
4. Patients who have any malignant or likely malignant Central Nervous System (CNS) lesion visible on CT.
5. Evidence of clinically significant immunosuppression such as primary immunodeficiency (e.g. severe combined immunodeficiency disease).
6. Clinically significant cardiac disease. Examples would include unstable coronary artery disease, myocardial infarction within 6 months or class III or IV American Heart Association criteria for heart disease.
7. Patients who are at high medical risk because of non-malignant systemic disease including those with uncontrolled cardiac or respiratory disease, or other serious medical or psychiatric disorders which, in the lead clinician's opinion, would not make the patient a good candidate for adoptive TIL therapy.
8. Severe and active autoimmune disease.
9. On concomitant treatment with other experimental drugs within 4 weeks of TIL harvesting.
10. Patients not considered likely to comply with required follow up.
11. Patients with severe allergies, history of anaphylaxis or known allergies to the administered drugs.
12. Patients who have received any prior adoptive cell therapy or organ transplant (including stem cells).
13. Patients who are pregnant or breast feeding should be excluded from pre-screening
14. Patients with any contraindications to any of the components of the study Non Investigational Medicinal Products (cyclophosphamide, fludarabine, Interleukin-2) will be excluded
15. Patents who have received live vaccines within 4 weeks prior to TIL therapy will be excluded

Inclusion for Main Study

-Patients are eligible to be included in the Main Study only if all of the following criteria, and the inclusion criteria listed in Section 1.3.1, apply:

1. Women with metastatic platinum resistant high-grade serous ovarian cancer (HGSOC) who have recurrent disease (platinum resistant defined as progressing within 6 months of last platinum-containing combination chemotherapy. patients must have received at least 1 line of prior platinum-containing combination chemotherapy and have completed at least 4 cycles of this treatment).
2. Informed consent to Main Study
3. Confirmation from Sponsor of successful TIL growth
4. Measurable disease (by Response Evaluation Criteria in Solid Tumors 1.1) on CT within 4 weeks of main study entry
5. Left ventricular ejection fraction >50% on Echocardiogram scan
6. Patients must be willing to practice a highly effective method of birth control during treatment and for four months after receiving the preparative regime if appropriate.
7. World Health Organisation (WHO) Performance Status of 0 or 1 (Appendix 3)
8. Age equal to or greater than 18 years
9. Life expectancy > 6 months
10. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the Pre-Screening or Main Study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
11. Seronegative for HIV antibody, Hep B antigen, Hep C antibody and syphilis
12. Haematological and biochemical indices

Exclusion for Main Study

1. Patients receiving day 1 of their last cycle of chemotherapy or targeted therapy less than four weeks prior to pre-conditioning chemotherapy.
2. Patients receiving systemic immunosuppressive therapy including steroids at doses higher than 10mg/day of prednisolone (or equivalent) within four weeks of commencing pre-conditioning chemotherapy (unless this is required briefly as anti-emetic prophylaxis for the treatments detailed in above point 1). Patients who require such therapies intermittently due to pre-existing disorders are also excluded.
3. Patients who have any malignant or likely malignant Central Nervous System (CNS) lesion visible on CT.
4. Evidence of any active significant infection.
5. Evidence of clinically significant immunosuppression such as primary immunodeficiency (e.g. severe combined immunodeficiency disease).
6. Clinically significant cardiac disease. Examples would include unstable coronary artery disease, myocardial infarction within 6 months or class III or IV American Heart Association criteria for heart disease.
7. Patients who are at high medical risk because of non-malignant systemic disease including those with uncontrolled cardiac or respiratory disease, or other serious medical or psychiatric disorders which, in the lead clinician's opinion, would not make the patient a good candidate for adoptive TIL therapy.
8. Severe and active autoimmune disease.
9. Receiving concomitant treatment with any other experimental drugs within 4 weeks of pre-conditioning chemotherapy. Patients receiving experimental immunotherapies will be discussed with the sponsor.
10. Patients not considered likely to comply with required follow up.
11. Patients with severe allergies, history of anaphylaxis or known allergies to the administered drugs.
12. Patients who are pregnant or breast feeding should be excluded from entering the study
13. Patients who have received any prior adoptive cell therapy or organ transplant (including stem cells).
14. Caution should be exercised for patients requiring regular drainage of ascites or pleural effusions. When there is sufficient fluid to be safely drained, drainage must be performed prior to trial enrolment and pre-conditioning chemotherapy in those patients.
15. Patients with any contraindications to any of the components of the study Non Investigational Medicinal Products (cyclophosphamide, fludarabine, Interleukin-2) will be excluded
16. Patents who have received live vaccines within 4 weeks prior to TIL therapy will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Sex of participants based on biological sex not self-representation as disease area being studied is Ovarian Cancer
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Disease objective response according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria | 6 weeks post treatment
  Subjects will have CT scan at 6 weeks post treatment to compare with baseline CT scans in order to assess disease response to therapy
Disease objective response according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria | 12weeks post treatment
  Subjects will have CT scan at 12 weeks post treatment to compare with baseline and previous post treatment CT scans in order to assess disease response to therapy
Disease objective response according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria | up to 24 months post treatment
  Subjects will have CT scan every 12 weeks after week 12 post treatment to compare with baseline and previous post treatment CT scans in order to assess disease response to therapy
Feasibility of treatment assessed by successful completion of planned treatment | 5 days post TIL therapy
  Subjects will receive lymphodepletion followed by a single TIL treatment and supportive IL-2
Tolerability and safety assessed according to NCI CTCAE v5.0 grading. | up to 24 months post TIL therapy
  Any adverse events related to study treatment will be recorded and assessed

SECONDARY OUTCOMES:
Percentage change in CA125 according to the Gynaecologic Cancer InterGroup CA125 response definition | up to 24 months post TIL therapy
  Serum level of CA125 will be measured in patients on day of discharge, 4weeks, 6weeks,12weeks and 3 monthly post TIL treatment
Feasibility assessed by successful completion of planned treatment. | 5 days post TIL therapy
  Subjects will receive lymphodepletion followed by a single TIL treatment and supportive IL-2
Progression free survival | up to 24 months post TIL therapy
  This will be measured by time from treatment initiation (from first day of pre-conditioning chemotherapy to radiological disease progression, relapse or death due to any cause
Duration of overall response and stable disease | up to 24 months post TIL therapy
  This is measured by time from response until radiological progression
Tolerability and safety assessed according to NCI CTCAE v5.0 grading | up to 24 months post TIL therapy
  Any adverse events related to study treatment will be recorded and assessed
Objective response by RECIST v1.1 | up to 24months post TIL therapy
  Subjects who have received CoTIL-01 will have CT scan at 6 weeks, 12 weeks, then very 12 weeks post treatment to compare with baseline and previous post treatment CT scans in order to assess disease response to therapy

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Thistlethwaite, PhD, MRCP, Principal Investigator — The Christie Hospital
Locations (2):
- United Kingdom (2):
  - Queens Elizabeth Hospital, Birmingham
  - The Christies Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No